CLINICAL TRIAL: NCT00249392
Title: Epidemiologic, Laboratory, and Clinical Characterization of Individuals With Ocular Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nanjing Medical University (Other)
Other Study IDs: ICP008
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Ocular Diseases
Keywords: ocular diseases; risk factors; genetic factors

SUMMARY:
Environmental and genetic factors may play a role in the progression of ocular diseases (cataract, retinopathy, age-related macular degeneration, glaucoma, retinal detachment, ocular tumor, etc.). The goal of this project is to establish a series of case-control studies to evaluate risk factors of ocular diseases in China.

DETAILED DESCRIPTION:
This study is designed to investigate the epidemiologic, genetic, laboratory and clinical characterization of individuals with ocular diseases (cataract, retinopathy, age-related macular degeneration, glaucoma, retinal detachment, ocular tumor, etc.). We will accrue approximately 800 patients as experimental group. The control group consists of age/sex frequency-matched subjects who will be confirmed without ocular diseases. We will explore the environmental (including family history, life style, diet, physical activity, neuropsychological functioning，plasma levels of oxidative stress and angiogenic factors, etc.) and genetic (including oxidative stress and angiogenic factors, etc.) risk factors. We will study the association between various environmental risk factors with the clinical characterization and correlation between the genetic polymorphisms and the presence of various ocular diseases.

ELIGIBILITY:
Inclusion Criteria:

* This is a study only of Chinese.
* Subjects will be allowed to participate if they self-identify as Chinese.
* Individuals with ocular diseases (cataract, retinopathy, age-related macular degeneration, glaucoma, retinal detachment, ocular tumor, etc.) will be allowed to participate. To participate in the study as the control, subjects should be confirmed without ocular diseases.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, Ph.D, Principal Investigator — Department of Pharmacology, Institute of Clinical Pharmacology, Nanjing Medical University
Locations (1):
- Department of Pharmacology, Institute of Clinical Pharmacology, Nanjing Medical University, Nanjing, Jiangsu, China